CLINICAL TRIAL: NCT01770509
Title: A Randomized, Parallel Group, Controlled Study to Assess the Efficacy and Safety of NMBM in the Treatment of Subjects With a Post-cellulitis and Venous Leg Ulcer
Brief Title: The Effect of the Cosmetic Cream NMBM on Leg Ulcers - a Pilot Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Lederman Consulting Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA -11- 9204-SG-CTIL
Record Dates: First submitted 2013-01-13; First posted 2013-01-17 (Estimated); Results first posted 2017-01-11 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2016-06

CONDITIONS: Ulcer; Venous Ulcer; Skin Ulcer; Leg Ulcer
Keywords: Chronic venous leg ulcers; Venous ulcer; Stasis ulcer; Varicose ulcer
MeSH Terms: conditions — Ulcer; Varicose Ulcer; Skin Ulcer; Leg Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of care (Active Comparator): Standard of care: Dressings +Compression garments
  Interventions: Other: Compression garments
- Application of NMBM (Experimental): Daily application of NMBM
  Interventions: Device: NMBM; Other: Compression garments

INTERVENTIONS:
Device: NMBM — Daily application of NMBM in addition to compression therapy
  Arms: Application of NMBM
Other: Compression garments — Compression garments

SUMMARY:
Ulcers of the lower extremities, caused by chronic venous insufficiency and cellulitis are common in patients older than 65 years and cause a significant morbidity.

Natural Matrix Bio polymer Membrane (NMBM) is a novel topical cosmetic cream containing a mix of natural waxes, sugars and lipids. The aim of this study is to test whether of Natural Matrix Bio polymer Membrane (NMBM) is effective as an adjunctive therapy to the treatment of venous stasis and post-erysipelas leg ulcers.

DETAILED DESCRIPTION:
Ulcers of the lower extremities, particularly in patients older than 65 years, are common among the population. Studies estimate the prevalence of current chronic leg ulcers at approximately 1%. The most common cause (approximately 80%) is thought to be chronic venous insufficiency disease. Recurrent cellulitis is an additional common cause. The ulcers cause a significant morbidity and negative impact on the patients' quality of life. The care of chronic vascular ulcers places a significant burden on the patient and the health care system. Additionally, these nonhealing ulcers place the patient at much higher risk for lower extremity amputation.

Natural Matrix Bio polymer Membrane (NMBM) is a novel topical cosmetic cream containing a mix of natural waxes, sugars and lipids. The aim of this study is to test whether of Natural Matrix Bio polymer Membrane (NMBM) is effective as an adjunctive therapy to the treatment of venous stasis and post-erysipelas leg ulcers.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated written Institutional Review Board (IRB) or Independent Ethics Committee (IEC) approved informed consent obtained from the subject in accordance with the local regulations;
2. Male or female subjects, ≥18 to ≤90 years of age
3. Patient with venous or predominantly venous leg ulcer (ankle-brachial index > 0.8)
4. Chronic venous insufficiency or post-erysipelas ulcer
5. Ulcer size between 5 and 170 sq cm, inclusive
6. Ulcer present for at least one month
7. ankle-brachial index >0.7

Exclusion Criteria:

1. Suffers from diabetes mellitus with HbA1c ≥ 8%
2. Albumin less than

2. 2. Patients with the following abnormal laboratory test levels hemoglobin <10.5 g/dL platelet count <100 x 109/L serum albumin level < 2.5 g/dL 3. Suffers from clinically significant arterial disease 34. Has a known allergy to any of the compounds that are part of this protocol 45. Has evidence of the ulcer and / or infection extending to the underlying muscle, tendon or bone 56. Has used any investigational drug(s) within 30 days preceding randomization 67. Is unable to manage self-treatment 78. Is pregnant, nursing mother or a woman of child bearing potential who is not using an adequate form of contraception (or abstinence) 8. 9. Suffers from a condition which in the opinion of the Investigator would compromise the safety of the subject and / or the quality of the data 9. 10. Unwilling or unable to comply with study requirements.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-02; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shoshana Greenberger, MD PhD, Principal Investigator — The Department of Dermatology, Sheba Medical Center
Locations (1):
- The Department of Dermatology, Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard of Care | Application of NMBM
Started | 12 | 17
Completed | 11 | 14
Not Completed | 1 | 3
Not completed — Injury | 0 | 1
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Application of NMBM | Total
Number analyzed (Participants) | 12 | 17 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.54 (7.7) | 68.17 (13.9) | 70.9 (12.6)
Gender [Count of Participants; unit: Participants]
  Female | 5 | 9 | 14
  Male | 7 | 8 | 15
Region of Enrollment [Number; unit: participants]
  Israel | 12 | 17 | 29

OUTCOME MEASURES:

1. Primary Outcome: Logarithm of Percentage of Baseline Ulcer Size
Description: Logarithm of percentage of baseline ulcer size. Log (ulcer area at 4 weeks/ulcer area at baseline *100) Ulcer area measured as longest ulcer length x longest ulcer width
Time Frame: From start of treatment to 4 weeks
Population: Analysis is based on measures from each ulcer, when some participants had more than one ulcer
Measure: Mean (Standard Deviation); unit: Mean of log (percentage of baseline area
Units Other Than Participants: Ulcers
Arm/Group | Standard of Care | Application of NMBM
Number analyzed (Participants) | 11 | 14
Number analyzed (Ulcers) | 17 | 19
Mean of log (percentage of baseline area | 3.6043 (2.16636) | 3.5030 (2.11130)
Statistical Analysis 1: Comparison: Standard of Care vs Application of NMBM; Test type: Superiority or Other; p = 0.652, ANOVA; General Linear Model ANOVA with repeated measures

2. Secondary Outcome: Alleviation of Pain
Description: Pain in week 4, assessed by the patient on a visual analogue pain score from 0 to 10. 0 represents no pain, 10 represents worst pain
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard of Care | Application of NMBM
Number analyzed (Participants) | 11 | 14
units on a scale | 2.45 (1.29) | 1.68 (1.62)
Statistical Analysis 1: Comparison: Standard of Care vs Application of NMBM; Test type: Superiority or Other; p = 0.645, ANOVA; General Linear Model ANOVA with repeated measures

3. Secondary Outcome: Incidence of Adverse Events at 4 Weeks
Description: Number of patients with adverse effects at 4 weeks
Time Frame: 4 weeks
Measure: Number; unit: Number of patients with adverse events
Arm/Group | Standard of Care | Application of NMBM
Number analyzed (Participants) | 11 | 14
Number of patients with adverse events | 1 | 3

4. Secondary Outcome: Incidence of Adverse Events
Description: Number of adverse effects at 4 weeks
Time Frame: 4 weeks
Measure: Number; unit: number of adverse effects
Arm/Group | Standard of Care | Application of NMBM
Number analyzed (Participants) | 11 | 14
number of adverse effects | 1 | 3

5. Secondary Outcome: Time to Complete Closure
Time Frame: 4 weeks
Population: Data was not collected as time to ulcer closure has been beyond the study period in the majority of patients
Arm/Group | Standard of Care | Application of NMBM
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Standard of Care | Application of NMBM
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/14
Other Adverse Events (participants affected / at risk) | 1/11 | 3/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard of Care (N=11) | Application of NMBM (N=14)
local irritation (Skin and subcutaneous tissue disorders) | 0 | 3 — Local erythema or burning
wound infection (Skin and subcutaneous tissue disorders) | 1 | 0 — Secondary infection of wound treated by antibiotics

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No